CLINICAL TRIAL: NCT01903395
Title: Nurse-led Colon Cancer Risk Counseling for First-degree Relatives to Enhance Use of Colonoscopy
Brief Title: Risk-adapted Screening in First-degree Relatives of Patients With Colorectal Cancer
Acronym: FAMKOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Alexander Bauer, PhD, Martin-Luther-Universität Halle-Wittenberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NKP332-032
Record Dates: First submitted 2013-07-11; First posted 2013-07-19 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal Neoplasms/*drug therapy/*secondary; Health Services Accessibility; Humans; Supportive Care Needs; Psychooncology; Primary Health Care/*methods; Treatment Outcome; Socioeconomic Factors; Quality Assurance, Health Care; Adult; Aged; Aged, 80 and over
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nurse-led counselling (Experimental): First-degree relatives of patients undergoing active treatment for colorectal cancer are offered a nurse-led counselling by telephone regarding emotional and cognitive barriers to screening utilization.
  Interventions: Behavioral: Nurse-led counselling
- Usual Care (No Intervention): Usual print media, offered standardly by the recruiting centres.

INTERVENTIONS:
Behavioral: Nurse-led counselling — Nurse-led telephone counselling to double the utilization of preventive colonoscopy
  Arms: Nurse-led counselling

SUMMARY:
BACKGROUND: First-degree relatives of patients with colorectal cancer are at increased risk for colorectal cancer as well. Nevertheless, participation in the German national screening program stagnates at 2-3 percent per year even in this high-risk population.

AIM: The study is aimed to increase the portion of the first-degree relatives on 50% which take up a preventive colonoscopy.

METHODS: Cluster-randomized controlled multi-center trial. Study sites (clusters) are mainly certified cancer centers and office-based gastroenterologists from all over Germany. Index-patients with colorectal cancer of different stages are asked to hand over the study material to their relatives, consisting of an invitation to a nurse-led counseling on preventive colonoscopy and an one-to-one appointment with a clinical expert of one of the study sites next.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 and over
* being first-degree relatives of patients with diagnosed colorectal cancer
* able to understand German

Exclusion Criteria:

* Familial Adenomatous Polyposis
* utilization of diagnostic colonoscopy within the past 5 years
* being ever treated for colorectal cancer
* actual inflammatory bowl disease
* comorbidities associated with reduced further life expectancy (ECOG performance status >3

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2012-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
utilization of preventive colonoscopy | utilization within 30 days after enrolement

SECONDARY OUTCOMES:
Rate of advanced adenomas or carcinomas in situ | Rate within 6 month after enrolement
post-operative complications associated with the colonoscopy | within 30 days after enrolement
barriers to the use of preventive colonoscopy | within 30 day after enrolement, additional at 6 months after enrolement
  Barriers against preventive colonoscopy are very common among the healthy population. Such barriers can bei either of cognitive (e.g. being afraid of the potential diagnosis) or emotional nature (e.g. shame to be exposed naked to the examiners).
  Barriers are assessed by Barriers Questionnaire-II (BQ-II) during telephone counselling.
effectiveness and cost-effectiveness of nurse-led counselling | within 30 days after enrolement
time delay between signed informed consent and utilization of colonoscopy | at utilization of the colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Bauer, PhD, Principal Investigator — Martin-Luther-University Halle-Wittenberg, Medical Faculty, Institute for Health and Nursing Science
Locations (33):
- Germany (33):
  - Kliniken Landkreis Sigmaringen GmbH, Sigmaringen, Baden-Wurttemberg
  - Klinikum Ludwigsburg, Ludwigsburg, Baden-Würtemberg
  - Diakoniekrankenhaus Mannheim, Mannheim, Baden-Würtemberg
  - Klinikum Stuttgart Krankenhaus Bad Cannstatt, Stuttgart, Baden-Würtemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Würtemberg
  - Klinikum Aschaffenburg, Aschaffenburg, Bavaria
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Stiftung Juliusspital Würzburg, Würzburg, Bavaria
  - Klinikum Barnim, Eberswalde, Brandenburg
  - Klinikum Hanau, Hanau, Hesse
  - Universitätsklinikum Gießen und Marburg, Marburg, Hesse
  - Städtisches Klinikum Braunschweig, Braunschweig, Lower Saxony
  - Allgemeines Krankenhaus Celle, Celle, Lower Saxony
  - Städtisches Klinikum Lüneburg, Lüneburg, Lower Saxony
  - Klinikum Osnabrück GmbH, Osnabrück, Lower Saxony
  - HELIOS Kliniken Schwerin, Schwerin, Mecklenburg-Vorpommern
  - Universitätsklinikum Knappschaftskrankenhaus Ruhr Universität Bochum, Bochum, Nordrhein-Wetsfalen
  - Krankenhaus Köln-Holweide, Cologne, North Rhine-Westphalia
  - Klinik Evang. Krankenhaus Kalk, Cologne, North Rhine-Westphalia
  - Johanniter-Krankenhaus Rheinhausen, Duisburg, North Rhine-Westphalia
  - Sankt Elisabeth Hospital Gütersloh, Gütersloh, North Rhine-Westphalia
  - Klinikum Lüdenscheid, Lüdenscheid, North Rhine-Westphalia
  - Krankenhaus St. Marienwörth, Bad Kreuznach, Rhineland-Palatinate
  - Diakonissen-Stiftungs-Krankenhaus Speyer, Speyer, Rhineland-Palatinate
  - Gastroenterologische Schwerpunktpraxis Völklingen, Völklingen, Saarland
  - Evangelisches Diakonissenkrankenhaus Leipzig gGmbH, Leipzig, Saxony
  - Diakonissenkrankenhaus Dessau gemeinnützige GmbH, Dessau, Saxony-Anhalt
  - Klinikum Magdeburg gemeinnützige GmbH, Magdeburg, Saxony-Anhalt
  - HELIOS Klinik Sangerhausen, Sangerhausen, Saxony-Anhalt
  - Evangelisches Krankenhaus Paul Gerhardt Stift, Wittenberg, Saxony-Anhalt
  - Praxis für Innere Medizin Dr. med. Regine Lange, Wittenberg, Saxony-Anhalt
  - Westküstenklinikum Heide, Heide, Schleswig-Holstein
  - Universitätsklinikum Jena, Jena, Thuringia